CLINICAL TRIAL: NCT01951638
Title: A Randomized Parallel-group, Placebo-controlled, Double-blind, Multi-center Dose Finding Phase II Trial Exploring the Pharmacodynamic Effects, Safety and Tolerability, and Pharmacokinetics of Four Dose Regimens of the Oral sGC Stimulator BAY1021189 Over 12 Weeks in Patients With Worsening Heart Failure and Preserved Ejection Fraction (HFpEF)
Brief Title: Phase IIb Safety and Efficacy Study of Four Dose Regimens of BAY1021189 in Patients With Heart Failure and Preserved Ejection Fraction Suffering From Worsening Chronic Heart Failure (SOCRATES-PRESERVED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15829; 2013-002288-25 (EudraCT Number)
Record Dates: First submitted 2013-09-24; First posted 2013-09-26 (Estimated); Results first posted 2021-02-12 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
Keywords: Worsening Heart Failure; Heart Failure with Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — vericiguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Vericiguat (BAY1021189)(10 mg) (Experimental): 2.5 mg orally once daily for 2 weeks, up-titration to 5 mg orally once daily for 2 weeks, up-titration to 10 mg orally once daily for 8 weeks
  Interventions: Drug: Vericiguat (BAY1021189) (1.25 mg); Drug: Vericiguat (BAY1021189) (5 mg)
- Vericiguat (BAY1021189) (5 mg) (Experimental): 2.5 mg orally once daily for 2 weeks, then 5 mg orally once daily for 10 weeks (with sham titration)
  Interventions: Drug: Vericiguat (BAY1021189) (1.25 mg); Drug: Vericiguat (BAY1021189) (5 mg)
- Vericiguat (BAY1021189) (2.5 mg) (Experimental): 2.5 mg orally once daily for 12 weeks (with sham titrations)
  Interventions: Drug: Vericiguat (BAY1021189) (1.25 mg)
- Vericiguat (BAY1021189) (1.25 mg) (Experimental): 1.25 mg orally once daily for 12 weeks (with sham titrations)
  Interventions: Drug: Vericiguat (BAY1021189) (1.25 mg)
- Placebo (Placebo Comparator): Orally once daily for 12 weeks (with sham titrations)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) (1.25 mg) — 1.25 mg BAY1021189 tablets
  Arms: Vericiguat (BAY1021189) (1.25 mg); Vericiguat (BAY1021189) (2.5 mg); Vericiguat (BAY1021189) (5 mg); Vericiguat (BAY1021189)(10 mg)
Drug: Vericiguat (BAY1021189) (5 mg) — 5 mg BAY1021189 tablets
  Arms: Vericiguat (BAY1021189) (5 mg); Vericiguat (BAY1021189)(10 mg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Objective of the study is to find the optimal dose of the once daily oral soluble guanylate cyclase stimulator (sGC) BAY1021189 for Phase III that can be given in addition to standard diuretic and comorbidity treatment for heart failure with preserved ejection fraction (HFpEF)

ELIGIBILITY:
Inclusion Criteria:

* Worsening chronic heart failure (WCHF) requiring hospitalization (or intravenous diuretic treatment for HF without hospitalization) with initiation of study treatment after clinical stabilization
* Left ventricular ejection fraction (LVEF) >/= 45% by echocardiography at randomization

Exclusion Criteria:

* Intravenous inotropes at any time after hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2013-11-06 (Actual); Primary Completion 2015-08-18 (Actual); Study Completion 2015-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (137):
- United States (17):
  - Fountain Valley, California
  - Fort Lauderdale, Florida
  - Naples, Florida
  - Macon, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Newark, New Jersey
  - Buffalo, New York
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Milwaukee, Wisconsin
- Australia (4):
  - Darlinghurst, New South Wales
  - Brisbane, Queensland
  - Redcliffe, Queensland
  - Hobart, Tasmania
- Austria (5):
  - Sankt Pölten, Lower Austria
  - Graz, Styria
  - Linz, Upper Austria
  - Salzburg
  - Vienna
- Belgium (8):
  - Bruges
  - Bruxelles - Brussel
  - Ghent
  - Gilly
  - Huy
  - Mechelen
  - Mol
  - Roeselare
- Bulgaria (3):
  - Burgas
  - Sofia
  - Stara Zagora
- Canada (5):
  - Toronto, Ontario
  - Montreal, Quebec
  - Saint-Jean-sur-Richelieu, Quebec
  - Sherbrooke, Quebec
  - Québec
- Czechia (2):
  - Kroměříž
  - Prague
- Denmark (3):
  - Aalborg
  - Holbæk
  - Randers
- France (4):
  - Bron
  - Pessac
  - Rouen
  - Toulouse
- Germany (10):
  - Bad Krozingen, Baden-Wurttemberg
  - München, Bavaria
  - Bad Homburg, Hesse
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Homburg, Saarland
  - Erfurt, Thuringia
  - Hamburg
- Greece (3):
  - Athens
  - Chaïdári
  - Nea Ionia / Athens
- Hungary (3):
  - Budapest
  - Kistarcsa
  - Székesfehérvár
- Israel (10):
  - Afula
  - Ashkelon
  - Hadera
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Rehovot
  - Tel Aviv
  - Tiberias
  - Zrifin
- Italy (6):
  - Bergamo, Lombardy
  - Brescia, Lombardy
  - Milan, Lombardy
  - Pavia, Lombardy
  - Ancona, The Marches
  - Arezzo, Tuscany
- Japan (22):
  - Iizuka, Fukuoka
  - Himeji, Hyōgo
  - Higashiibaraki, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Takamatsu, Kagawa-ken
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Uji, Kyoto
  - Naha, Okinawa
  - Sakai, Osaka
  - Takatsuki, Osaka
  - Komatsushimachō, Tokushima
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Fukui
  - Hiroshima
  - Kumamoto
  - Nagasaki
  - Osaka
  - Tokushima
  - Toyama
- Netherlands (4):
  - Amsterdam
  - Heerenveen
  - Leeuwarden
  - Sneek
- Poland (6):
  - Bialystok
  - Krakow
  - Lodz
  - Olsztyn
  - Poznan
  - Szczecin
- Portugal (2):
  - Almada
  - Lisbon
- Singapore, Singapore
- Seoul, South Korea
- Spain (5):
  - Santander, Cantabria
  - Majadahonda, Madrid
  - El Palmar, Murcia
  - Barcelona
  - Valencia
- Sweden (5):
  - Helsingborg
  - Karlstad
  - Linköping
  - Örebro
  - Stockholm
- Switzerland (2):
  - Lugano, Canton Ticino
  - Geneva
- Taiwan (4):
  - Kaohsiung City
  - New Taipei City
  - Taipei
  - Taoyuan District
- United Kingdom (2):
  - Chesterfield, Derbyshire
  - Stevenage, Hertfordshire

REFERENCES:
- [Background] Pieske B, Butler J, Filippatos G, Lam C, Maggioni AP, Ponikowski P, Shah S, Solomon S, Kraigher-Krainer E, Samano ET, Scalise AV, Muller K, Roessig L, Gheorghiade M; SOCRATES Investigators and Coordinators. Rationale and design of the SOluble guanylate Cyclase stimulatoR in heArT failurE Studies (SOCRATES). Eur J Heart Fail. 2014 Sep;16(9):1026-38. doi: 10.1002/ejhf.135. Epub 2014 Jul 24. PMID 25056511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 158 centers in 25 countries between 06 November 2013 (first subject first visit) and 16 September 2015 (last subject last visit).
Pre-assignment Details: Overall, 632 subjects were enrolled, of them 477 were randomized and 475 were treated. Among the 477 subjects who were randomized, 404 subjects completed both treatment and follow-up [FU] periods. All arms in FU period were mutually exclusive, this question below is ticked No because of database validation rule constraints.
Groups:
- Placebo: Subjects received placebo matched to vericiguat (BAY1021189) orally once daily for 12 weeks. Sham titrations included on Days 14 and 28.
- BAY1021189 1.25 mg: Subjects received vericiguat (Verquvo, BAY1021189) 1.25 milligram (mg) orally once daily for 12 weeks. Sham titrations included on Days 14 and 28.
- BAY1021189 2.5 mg: Subjects received vericiguat (Verquvo, BAY1021189) 2.5 mg orally once daily for 12 weeks. Sham titrations included on Days 14 and 28.
- BAY1021189 2.5 mg to 5 mg: Subjects received vericiguat (Verquvo, BAY1021189) for 12 weeks, starting on 2.5 mg once daily with potential up-titration to 5 mg after 14 or 28 days. Sham titration included on Day 28.
- BAY1021189 2.5 mg to 10 mg: Subjects received vericiguat (Verquvo, BAY1021189) for 12 weeks, starting on 2.5 mg once daily with potential up-titration to 5 mg once daily after 14 days, and up-titration to 10 mg once daily after 28 days.
Period: Treatment Period
Arm/Group | Placebo | BAY1021189 1.25 mg | BAY1021189 2.5 mg | BAY1021189 2.5 mg to 5 mg | BAY1021189 2.5 mg to 10 mg
Started | 93 | 96 | 96 | 96 | 96
Completed | 80 | 82 | 83 | 80 | 86
Not Completed | 13 | 14 | 13 | 16 | 10
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 0
Not completed — Protocol-driven decision point | 1 | 3 | 0 | 0 | 0
Not completed — Logistical difficulties | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 6 | 4 | 5 | 4
Not completed — Death | 0 | 0 | 0 | 3 | 1
Not completed — Adverse Event | 3 | 4 | 8 | 6 | 5
Period: Follow-up Period
Arm/Group | Placebo | BAY1021189 1.25 mg | BAY1021189 2.5 mg | BAY1021189 2.5 mg to 5 mg | BAY1021189 2.5 mg to 10 mg
Started | 89 | 95 | 95 | 88 | 94
Completed | 87 | 86 | 90 | 80 | 89
Not Completed | 2 | 9 | 5 | 8 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Logistical difficulties | 0 | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 5 | 2 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 1 | 4 | 1
Not completed — Adverse Event | 0 | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BAY1021189 1.25 mg | Placebo | BAY1021189 2.5 mg | BAY1021189 2.5 mg to 5 mg | BAY1021189 2.5 mg to 10 mg | Total
Number analyzed (Participants) | 96 | 93 | 96 | 96 | 96 | 477
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (10) | 73.7 (9.1) | 72 (10.7) | 73.9 (7.9) | 72.5 (10.2) | 73.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 46 | 43 | 43 | 44 | 227
  Male | 45 | 47 | 53 | 53 | 52 | 250

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Log-transformed N-terminal Pro-brain Natriuretic Peptide (NT-proBNP)
Description: NTproBNP is a circulating plasma biomarker of cardiovascular function and prognosis in heart failure (HF).
Time Frame: Baseline, Week 12 (end of treatment [EOT])
Population: Per Protocol Set (PPS) NT-pro BNP: included all subjects randomized to treatment who had a valid measurement of NT-pro BNP at baseline and at Week 12 (Visit 5) and showed no major protocol deviations.
Measure: Mean (Standard Deviation); unit: log-transformed picograms per milliliter
Arm/Group | Placebo | BAY1021189 1.25 mg | BAY1021189 2.5 mg | BAY1021189 2.5 mg to 5 mg | BAY1021189 2.5 mg to 10 mg
Number analyzed (Participants) | 73 | 77 | 78 | 57 | 60
log-transformed picograms per milliliter | -0.098 (0.778) | -0.047 (0.788) | 0.071 (0.818) | 0.057 (0.819) | -0.023 (0.705)
Statistical Analysis 1: Comparison: Placebo; For the primary analysis, the three highest active treatment groups BAY1021189 (2.5mg, 2.5 to 5mg, 2.5 to 10mg) were pooled and compared to the assigned placebo treatment group with a one-sided two-sample t-test. The Hochberg procedure was used to test the two primary end points at study-wise significance level of 5%. Results are reported including 90% confidence intervals (CI) for the difference of means. The difference between the comparison groups is difference of means on the log scale; Test type: Other; p = 0.8991, t-test, 1 sided; Log-Scale mean difference = 0.137, 90% CI 2-sided [-0.04 to 0.31]
Statistical Analysis 2: Comparison: Placebo vs BAY1021189 2.5 mg to 10 mg; Pairwise comparisons to placebo were performed in a hierarchical manner (from BAY1021189 from 2.5 to 10mg dose arm to BAY1021189 1.25mg dose arm). In accordance with the specification in the protocol these secondary analyses are considered exploratory only, since the primary analyses were not significant; Test type: Other; p = 0.7194, t-test, 1 sided; Log-Scale mean difference = 0.076, 95% CI 2-sided [-0.18 to 0.33]
Statistical Analysis 3: Comparison: Placebo vs BAY1021189 2.5 mg to 5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.8653, t-test, 1 sided; Log-Scale mean difference = 0.156, 95% CI 2-sided [-0.12 to 0.43]
Statistical Analysis 4: Comparison: Placebo vs BAY1021189 2.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.9041, t-test, 1 sided; Log-Scale mean difference = 0.171, 95% CI 2-sided [-0.09 to 0.43]
Statistical Analysis 5: Comparison: Placebo vs BAY1021189 1.25 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.6572, t-test, 1 sided; Log-Scale mean difference = 0.052, 95% CI 2-sided [-0.2 to 0.3]

2. Primary Outcome: Change From Baseline to Week 12 in Left Atrial Volume (LAV)
Description: Left atrial volume was measured by echocardiography.
Time Frame: Baseline, Week 12 (EOT)
Population: PPS Left Atrial Volume (LAV) included all subjects randomized to treatment who had a valid measurement of LAV at baseline and at Week 12 (Visit 5) and showed no major protocol deviations.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Placebo | BAY1021189 1.25 mg | BAY1021189 2.5 mg | BAY1021189 2.5 mg to 5 mg | BAY1021189 2.5 mg to 10 mg
Number analyzed (Participants) | 67 | 77 | 78 | 57 | 59
milliliter | -3.361 (12.654) [lower limit 12.654] | -2.163 (7.895) [lower limit 7.895] | -2.142 (11.931) [lower limit 11.931] | -1.252 (16.139) [lower limit 16.139] | -1.654 (10.245) [lower limit 10.245]
Statistical Analysis 1: Comparison: Placebo; For the primary analysis, the three highest active treatment groups (BAY1021189 2.5mg, BAY1021189 2.5 to 5mg, BAY1021189 2.5 to 10mg) were pooled and compared to the assigned placebo treatment group with a one-sided two-sample t-test. The Hochberg procedure was used to test the two primary end points at study-wise significance level of 5%. Results are reported including 90% confidence intervals (CI) for the difference of means; Test type: Other; p = 0.8156, t-test, 1 sided; Mean Difference (Net) = 1.629, 90% CI 2-sided [-1.36 to 4.62]
Statistical Analysis 2: Comparison: Placebo vs BAY1021189 2.5 mg to 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.7945, t-test, 1 sided; Mean Difference (Net) = 1.707, 95% CI 2-sided [-2.39 to 5.8]
Statistical Analysis 3: Comparison: Placebo vs BAY1021189 2.5 mg to 5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.7917, t-test, 1 sided; Mean Difference (Net) = 2.109, 95% CI 2-sided [-3.01 to 7.23]
Statistical Analysis 4: Comparison: Placebo vs BAY1021189 2.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.7241, t-test, 1 sided; Mean Difference (Net) = 1.219, 95% CI 2-sided [-2.82 to 5.26]
Statistical Analysis 5: Comparison: Placebo vs BAY1021189 1.25 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.7546, t-test, 1 sided; Mean Difference (Net) = 1.198, 95% CI 2-sided [-2.23 to 4.63]

3. Other Pre Specified Outcome: Change From Baseline to Week 12 Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured after at least 10 minutes resting in a sitting position (3 measurements taken approximately 2 minutes apart).The changes in blood pressure were recorded and the mean of the three measurements was analyzed.
Time Frame: Baseline, Week 12 (EOT)
Population: Safety Analysis Set (SAF) with evaluable subjects for this endpoint.
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Placebo | BAY1021189 1.25 mg | BAY1021189 2.5 mg | BAY1021189 2.5 mg to 5 mg | BAY1021189 2.5 mg to 10 mg
Number analyzed (Participants) | 80 | 82 | 83 | 61 | 61
millimeter of mercury
  Change in SBP | 1.458 (18.865) | 0.703 (16.993) | -1.819 (19.438) | -1.486 (17.179) | -0.913 (15.498)
  Change in DBP | 1.887 (11.435) | 0.911 (10.037) | -2.173 (11.249) | -1.142 (11.4) | -0.629 (10.271)

4. Other Pre Specified Outcome: Change From Baseline to Week 12 in Heart Rate
Description: Heart rate was measured after 10 minutes resting in a sitting position (3 measurements taken approximatly 2 minutes apart). The changes in heart rate were recorded and the mean of the three measurements was analyzed.
Time Frame: Baseline, Week 12 (EOT)
Population: Safety Analysis Set (SAF) with evaluable subjects for this endpoint.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | BAY1021189 1.25 mg | BAY1021189 2.5 mg | BAY1021189 2.5 mg to 5 mg | BAY1021189 2.5 mg to 10 mg
Number analyzed (Participants) | 80 | 82 | 83 | 61 | 61
beats per minute | 3.287 (13.582) [lower limit 13.582] | 1.776 (11.42) [lower limit 11.42] | -0.373 (9.845) [lower limit 9.845] | 1.055 (13.331) [lower limit 13.331] | -2.623 (9.639) [lower limit 9.639]

5. Other Pre Specified Outcome: Number of Subjects With Clinical Events (Heart Failure Hospitalization and Cardio-vascular [CV] Mortality)
Description: Clinical events (heart failure and mortality) were analyzed as CV death, and HF hospitalization at specified time points.
Time Frame: Baseline up to Week 16 including 12 week treatment period and 4 week follow-up period
Population: Full Analysis Set (FAS) included all subjects who were randomized to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BAY1021189 1.25 mg | BAY1021189 2.5 mg | BAY1021189 2.5 mg to 5 mg | BAY1021189 2.5 mg to 10 mg
Number analyzed (Participants) | 93 | 96 | 96 | 96 | 96
Participants
  HF hospitalizations | 8 | 6 | 11 | 8 | 5
  CV Mortality | 1 | 0 | 0 | 5 | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were collected after first application of study medication up to 5 calendar days after end of treatment with study medication
Groups:
- BAY1021189 From 2.5 to 5 mg: Subjects received vericiguat (Verquvo, BAY1021189) for 12 weeks, starting on 2.5 mg once daily with potential up-titration to 5 mg once daily after 14 or 28 days. Sham titration included on Day 28.
- BAY1021189 From 2.5 to 10 mg: Subjects received vericiguat (Verquvo, BAY1021189) for 12 weeks, starting on 2.5 mg once daily with potential up-titration to 5 mg once daily after 14 days, and up-titration to 10 mg once daily after 28 days.
Arm/Group | Placebo | BAY1021189 1.25 mg | BAY1021189 2.5 mg | BAY1021189 From 2.5 to 5 mg | BAY1021189 From 2.5 to 10 mg
All-Cause Mortality (participants affected / at risk) | 1/93 | 0/96 | 1/95 | 7/95 | 2/96
Serious Adverse Events (participants affected / at risk) | 20/93 | 20/96 | 24/95 | 18/95 | 21/96
Other Adverse Events (participants affected / at risk) | 21/93 | 33/96 | 40/95 | 38/95 | 33/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=93) | BAY1021189 1.25 mg (N=96) | BAY1021189 2.5 mg (N=95) | BAY1021189 From 2.5 to 5 mg (N=95) | BAY1021189 From 2.5 to 10 mg (N=96)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 6 (6) | 4 (4) | 7 (12) | 5 (8) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 2 (3) | 4 (4) | 3 (3) | 2 (2) | 4 (5)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coagulation time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cervicogenic headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=93) | BAY1021189 1.25 mg (N=96) | BAY1021189 2.5 mg (N=95) | BAY1021189 From 2.5 to 5 mg (N=95) | BAY1021189 From 2.5 to 10 mg (N=96)
Cardiac failure (Cardiac disorders) | 5 (5) | 1 (1) | 3 (4) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (5) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (5) | 5 (5) | 4 (5)
Fatigue (General disorders) | 2 (3) | 2 (2) | 3 (3) | 6 (6) | 4 (4)
Oedema peripheral (General disorders) | 2 (3) | 3 (4) | 2 (3) | 6 (7) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 6 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 6 (8) | 1 (1) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 2 (2) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 2 (4) | 10 (11) | 6 (6) | 7 (7)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 6 (6) | 4 (4) | 4 (4)
Renal failure (Renal and urinary disorders) | 2 (3) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 6 (6) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7) | 9 (10) | 5 (6) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 4 (4) | 4 (6) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
End points, "Health-related quality of life, Composite Congestion Score, NYHA function class, echo parameters other than LAV, biomarker and background HF therapies" were exploratory. "Incidence of atrial fibrillation" is reported in AE section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No